CLINICAL TRIAL: NCT05843487
Title: Association Between Carotid Plaque Length and Cardiovascular Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Yueyang Hospital, Shanghai University of Traditional Chinese medicine (Unknown); Putuo Hospital, Shanghai University of Traditional Chinese Medicine (Unknown); 904th Hospital of the Joint Logistics Support Force of the PLA (Other); Gongli Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CPL
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease; Carotid Plaque
Keywords: Carotid Artery Ultrasound; Carotid Plaque; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid plaque length: Patients underwent carotid ultrasonography and first coronary angiography simultaneously

SUMMARY:
This multicenter study involved 5 hospitals (Changhai Hospital; Yueyang Hospital of Shanghai University of Traditional Chinese Medicine; Gongli Hospital; Putuo Hospital of Shanghai University of Traditional Chinese Medicine; No. 904 Hospital of the PLA Joint Logistics Support Force Wuxi). The study enrolled 5000 consecutive patients without known CAD who underwent first coronary angiography for stable chest pain and carotid ultrasound was performed during hospitalization from January 2017 through December 2018.

DETAILED DESCRIPTION:
Patients who had obstructive CAD (defined as ≥50% luminal stenosis) confirmed by coronary angiography and who underwent carotid scanning were included in the final analysis.Carotid ultrasonography was performed simultaneously, and carotid intima-media thickness (IMT), maximum thickness and length of all plaques were measured.The incidence of major adverse cardiovascular events was recorded during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent coronary angiography for stable chest pain and carotid ultrasound simultaneously;
* Patients with obstructive CAD (≥50% coronary stenosis);

Exclusion Criteria:

* <18 years of age;
* previous carotid surgery or significant carotid artery disease;
* prior stroke or transient ischemic attack;
* previously documented CAD (including history of myocardial infarction, acute coronary syndrome, or coronary revascularization);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients without known CAD who underwent first coronary angiography for stable chest pain and carotid ultrasound was performed during hospitalization.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 3 years
  cardiovascular death, myocardial infarction, ischemic stroke and coronary revascularization

SECONDARY OUTCOMES:
all-cause death | 3 years
cardiovascular death | 3 years
myocardial infarction | 3 years
ischemic stroke | 3 years
coronary artery revascularization | 3 years
heart failure | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pan Li, PhD, Principal Investigator — Changhai Hospital; Jian Jian Na, MD, Study Director — Putuo Hospital; Liang Chen, MD, Study Director — 904th Hospital of the Joint Logistics Support Force of the PLA; Wei Zhang, MD, Study Director — Gongli Hospital; Yawei Yang, MD, Study Director — Yueyang Hospital
Locations (5):
- China (5):
  - No. 904 Hospital of the PLA Joint Logistics Support Force, Wuxi, Jiangsu
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Gongli Hospital, Shanghai, Shanghai Municipality
  - Putuo Hospital, Shanghai, Shanghai Municipality
  - Yueyang Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided